CLINICAL TRIAL: NCT04991181
Title: An Open-label Study to Assess the Absorption, Distribution, Metabolism and Excretion, Including the Mass Balance, of [14C] Labeled BIA 5-1058 and Metabolites Following a Single Oral Dose Administration in Healthy Male Subjects
Brief Title: Absorption, Distribution, Metabolism and Excretion of BIA 5-1058
Acronym: ADME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-51058-104; 2015-002407-28 (EudraCT Number)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — zamicastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIA 5-1058 (Experimental): Capsules; 400 mg; single dose; oral administration.
  Interventions: Drug: 400 mg BIA 5-1058

INTERVENTIONS:
Drug: 400 mg BIA 5-1058 — Capsules, oral administered to subjects between 08:00 and 09:00 hours in the morning of Day 1after an overnight fast of at least 10 hours. The study drug was swallowed together with 240 mL tap water (room temperature).
  Other Names: Zamicastat

SUMMARY:
the purpose of this study is:

* to determine the rate and routes of excretion of BIA 5-1058 and the mass balance in urine, feces and exhaled air, after a single oral dose of 400 mg 14C labeled BIA 5 1058 containing 3.7 Megabecquerel (MBq) of radiocarbon;
* to determine the pharmacokinetics (PK) of total radioactivity (TRA) in plasma and whole blood and to assess the blood-to-plasma ratio;
* to determine the PK of BIA 5-1058 and its metabolites in plasma.

DETAILED DESCRIPTION:
This was a Phase 1, single-center, open-label, absorption, distribution, metabolism, and excretion study in 8 healthy adult male subjects. Subjects received a single oral dose of 400 mg BIA 5-1058, containing approximately 3.7 MBq (0.08 milliSievert [mSv]) of 14C-BIA 5-1058 as oral capsules. Screening was between Day -21 and Day -2 and confinement period was of one period in the clinic involving drug administration on Day 1, with admission on Day 1 and discharge on Day 15 (336 hours post-dose).

ELIGIBILITY:
Inclusion Criteria:

1. Gender :male
2. Age :18-65 years, inclusive
3. Body Mass Index (BMI) :18.0-30.0 kg/m2 (BMI [kg/m2] = Body weight [kg] ÷ Height2 [m2]) at screening
4. Subjects, if not surgically sterilized, were willing to use adequate contraception and not donate sperm from admission to the clinical research center until 90 days after discharge on Day 15. Adequate contraception for the male subject (and his female partner) was defined as using hormonal contraceptives or an intrauterine device combined with at least 1 of the following forms of contraception: a diaphragm or cervical cap, or a condom. Also, total abstinence, in accordance with the lifestyle of the volunteer, was acceptable
5. All prescribed medication had to be stopped at least 30 days prior to admission to the clinical research center
6. All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (e.g., St. John's Wort) had to be stopped at least 14 days prior to admission to the clinical research center. An exception was made for paracetamol, which was allowed up to admission to the clinical research center
7. Ability and willingness to abstain from alcohol, methylxanthine-containing beverages or food (coffee, tea, cola, chocolate and "powerdrinks"), commercially available orange juice (because of a potential interaction of radioactivity and vitamin C), grapefruit (juice) and tobacco products from 48 hours prior to admission to in the clinical research center until discharge (Day 15)
8. Normal resting supine blood pressure and pulse showing no clinically relevant deviations as judged by the PI
9. Computerized (12-lead) ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the PI
10. All values for clinical laboratory tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the PI
11. Willing and able to sign the ICF.

Exclusion Criteria:

1. Employee of PRA or the Sponsor
2. Evidence of clinically relevant pathology or a medical history of a major pathology as judged by the PI
3. Frequent headaches and/or migraine, recurrent nausea, and/or vomiting (more than twice a month)
4. Mental handicap (i.e. a general or specific intellectual disability, resulting directly or indirectly from injury to the brain or from abnormal neurological development)
5. History of relevant drug and/or food allergies
6. Smoking more than 5 cigarettes, 1 cigar or 1 pipe daily; the use of tobacco products in the 48 hours (2 days) prior to admission to the clinical research center on Day 1 was not allowed
7. History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
8. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants and alcohol)
9. Average intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
10. Positive screen for hepatitis B surface antigen (HBsAg), anti hepatitis C virus (HCV) antibodies or anti human immunodeficiency virus (HIV) 1 and 2 antibodies
11. Participation in a drug study within 90 days prior to drug administration in the current study. Participation in more than 2 other drug studies in the 12 months prior to drug administration in the current study
12. Donation or loss of more than 100 mL of blood within 90 days prior to drug administration. Donation or loss of more than 1.5 liters of blood in the 10 months prior to drug administration in the current study
13. Subject with irregular bowel habits (more than 3 times a day or less than once every 2 days)
14. Strenuous exercise within 96 hours (4 days) prior to admission to the clinical research center
15. Significant and/or acute illness within 5 days prior to drug administration that may impact the safety of the subject, in the opinion of the PI
16. Participation in another ADME study with a radiation burden >0.1 mSv in the period of 1 year prior to screening
17. Exposure to radiation for diagnostic reasons (except dental X rays and plain X rays of thorax and bony skeleton [excluding spinal column]), during work or during participation in a clinical study in the period of 1 year prior to screening
18. Previous use of BIA 5 1058.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — healthy male subjects
Enrollment: 15 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Cmax - Maximum observed plasma concentration | Up to 20 days
  Pharmacokinetic Parameters for BIA 5-1058 (and Metabolites) in Plasma and for TRA in Plasma and Whole Blood.
  Blood sampling was collected at pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 120, 168, 240 and 336 hours post-dose, and at 504 (±24 h), 672 (±24 h), 1008 (±48 h), 1344 (±48 h), and 1848 (±72 h) hours post-dose
Tmax - Time to attain maximum observed plasma concentration | Up to 20 days
  Pharmacokinetic Parameters for BIA 5-1058 (and Metabolites) in Plasma and for TRA in Plasma and Whole Blood.
  Blood sampling was collected at pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 120, 168, 240 and 336 hours post-dose, and at 504 (±24 h), 672 (±24 h), 1008 (±48 h), 1344 (±48 h), and 1848 (±72 h) hours post-dose
AUC0-t Area under the plasma concentration-time curve up to time t, where t is the last point with concentrations above the lower limit of quantitation (LLOQ) | Up to 20 days
  Pharmacokinetic Parameters for BIA 5-1058 (and Metabolites) in Plasma and for TRA in Plasma and Whole Blood.
  Blood sampling was collected at pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 120, 168, 240 and 336 hours post-dose, and at 504 (±24 h), 672 (±24 h), 1008 (±48 h), 1344 (±48 h), and 1848 (±72 h) hours post-dose
AUC0-inf - Area under the plasma concentration-time curve from time 0 extrapolated to infinity | Up to 20 days
  Pharmacokinetic Parameters for BIA 5-1058 (and Metabolites) in Plasma and for TRA in Plasma and Whole Blood.
  Blood sampling was collected at pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 120, 168, 240 and 336 hours post-dose, and at 504 (±24 h), 672 (±24 h), 1008 (±48 h), 1344 (±48 h), and 1848 (±72 h) hours post-dose
t1/2 - Elimination half-life | Up to 20 days
  Pharmacokinetic Parameters for BIA 5-1058 (and Metabolites) in Plasma and for TRA in Plasma and Whole Blood.
  Blood sampling was collected at pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 120, 168, 240 and 336 hours post-dose, and at 504 (±24 h), 672 (±24 h), 1008 (±48 h), 1344 (±48 h), and 1848 (±72 h) hours post-dose
CLR - Renal clearance | Up to 20 days
  Pharmacokinetic Parameters for BIA 5-1058 (and Metabolites) in Plasma and for TRA in Plasma and Whole Blood.
  Blood sampling was collected at pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 120, 168, 240 and 336 hours post-dose, and at 504 (±24 h), 672 (±24 h), 1008 (±48 h), 1344 (±48 h), and 1848 (±72 h) hours post-dose
Aeurine - Cumulative amount excreted in urine | Up to 20 days
  Cumulative Recovery of Radioactivity in Urine URINE collection was at pre-dose (collected within 24 hours prior to drug administration) and at collection intervals of 0-6, 6-12, 12-24 and 24-48 hours post-dose, and in 24-hour collections intervals thereafter until discharge from the clinic on Day 15 (336 hours post-dose); and 24 hour collections on Days 21/22, 28/29, 42/43, 56/57 and 77/78, depending on recovery limits as assessed initially after Day 15.).
Ae feces - Cumulative amount excreted in feces | Up to 20 days
  Cumulative Recovery of Radioactivity in Feces
  FECES collection was at pre-dose and at collection intervals of 0-24, 24-48, 48 72, 72 96, 96 120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264, 264-288, 288-312 and 312-336 hours post-dose; and 24-hour collections on Days 21/22, 28/29, 42/43, 56/57 and 77/78, depending on recovery limits as assessed initially after Day. The pre dose sample was collected within 48 hours prior to drug administration (if collected at home before admission on Day 1, subjects recorded the time of collection and brought the sample at admission). From 48 h before returning to the clinic for the 24-hour collections, the subjects also collected stools at home and recorded the time of collection.
Aeair - Cumulative amount excreted in exhaled air | Up to 20 days
  Cumulative Recovery of Radioactivity in Exhaled Air.
  EXHALED AIR sampling was at pre-dose and 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168 and 240 hours post dose (with possible extension at 336 hours post-dose, if needed).
Aetotal - Total amount excreted, calculated as Aeurine + Aefeces + Aeair | Up to 20 days
  Cumulative Recovery of Radioactivity in Urine, Feces, Exhaled Air. URINE collection was at pre-dose (collected within 24 hours prior to drug administration) and at collection intervals of 0-6, 6-12, 12-24 and 24-48 hours post-dose, and in 24-hour collections intervals thereafter until discharge from the clinic on Day 15 (336 hours post-dose); and 24 hour collections on Days 21/22, 28/29, 42/43, 56/57 and 77/78, depending on recovery limits as assessed initially after Day 15.
  FECES collection was at pre-dose and at collection intervals of 0-24, 24-48, 48 72, 72 96, 96 120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264, 264-288, 288-312 and 312-336 hours post-dose; and 24-hour collections on Days 21/22, 28/29, 42/43, 56/57 and 77/78, depending on recovery limits as assessed initially after Day.
  EXHALED AIR sampling was at pre-dose and 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168 and 240 hours post dose (with possible extension at 336 hours post-dose, if needed).
TRA t1/2 plasma | Up to 20 days
  Excretion Rates of TRA in Plasma PLASMA Blood sampling was collected at pre-dose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 16, 24, 36, 48, 72, 120, 168, 240 and 336 hours post-dose, and at 504 (±24 h), 672 (±24 h), 1008 (±48 h), 1344 (±48 h), and 1848 (±72 h) hours post-dose
TRA t1/2 urine | Up to 20 days
  Excretion Rates of TRA in Urine
  URINE collection was at pre-dose (collected within 24 hours prior to drug administration) and at collection intervals of 0-6, 6-12, 12-24 and 24-48 hours post-dose, and in 24-hour collections intervals thereafter until discharge from the clinic on Day 15 (336 hours post-dose); and 24 hour collections on Days 21/22, 28/29, 42/43, 56/57 and 77/78, depending on recovery limits as assessed initially after Day 15
TRA t1/2 feces | Up to 20 days
  Excretion Rates of TRA in Feces
  FECES collection was at pre-dose and at collection intervals of 0-24, 24-48, 48 72, 72 96, 96 120, 120-144, 144-168, 168-192, 192-216, 216-240, 240-264, 264-288, 288-312 and 312-336 hours post-dose; and 24-hour collections on Days 21/22, 28/29, 42/43, 56/57 and 77/78, depending on recovery limits as assessed initially after Day. The pre dose sample was collected within 48 hours prior to drug administration (if collected at home before admission on Day 1, subjects recorded the time of collection and brought the sample at admission). From 48 h before returning to the clinic for the 24-hour collections, the subjects also collected stools at home and recorded the time of collection.

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences (PRA) - Early Development Services (EDS), Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided